CLINICAL TRIAL: NCT02934022
Title: Adding Maraviroc to the HAART Regimen of HIV-infected Patients Who Are Well Controlled, and the Effect on CD4 Lymphocyte Counts
Brief Title: Adding Maraviroc to the HAART Regimen of Well Controlled HIV-infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern California Institute for Research and Education (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WS719742
Record Dates: First submitted 2012-06-04; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: HIV Infection
Keywords: Maraviroc; HAART regimen; Immunologic response
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Maraviroc (Other)
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — 150 mg tablets, two or 4 tablets once daily (dependent upon concommitant medications)
  Other Names: Selzentry

SUMMARY:
Many patients on Highly Active Antiretroviral Therapy (HAART) are able to achieve a sustained response with viral loads becoming undetectable and staying undetectable, but do not have an increase in their CD4 counts to levels greater than 500. Adding maraviroc to the treatment regimen of these patients may result in an increase in their CD4 counts. As the patient would be continuing their prior regimen, they will likely continue with full control of viral replication.

DETAILED DESCRIPTION:
This is a prospective, open-label, non-controlled, non-randomized, single center study of the effect of adding the antiretroviral Maraviroc to the antiretroviral treatment regimen (HAART)of patients who have achieved a sustained virologic response to HAART but have had a sub-adequate immunologic response to treatment. Patients who have had a full virologic response (as defined by HIV-1 viral loads of < 48 copies/mL) for 12 months or more are defined as having a sub-adequate immunologic response if their CD4 lymphocyte count has not gone above 500.

This pilot study will contain up to 30 patients who will be followed over a period of 12 months starting from the date of enrollment and addition of maraviroc to their current highly active antiretroviral therapy regimen. The main outcome to be followed is the CD4 lymphocyte counts at baseline and after 12 months of treatment with the addition of maraviroc.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 positive.
2. Receiving highly active antiretroviral therapy (HAART).
3. HIV-1 viral load of < 48 copies for 12 months or more.
4. CD4 lymphocyte count that has not gone above 500. -

Exclusion Criteria:

1. Severe hepatic impairment (cirrhosis) or active Hepatitis C with liver transaminases > 5 times normal.
2. Severe renal impairment (creatinine clearance < 30 ml/min) or end-stage renal disease (ESRD) who are taking potent CYP3A4 inhibitors or inducers.
3. Receiving certain necessary medications that have the potential for serious drug-drug interactions with maraviroc. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in absolute CD4 lymphocyte count after addition of maraviroc for 12 months to the subject's current highly active antiretroviral therapy (HAART) regimen. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M. Berman, MD, PhD, Principal Investigator — VA Long Beach Healthcare System
Locations (1):
- VA Long Beach Healthcare System, Long Beach, California, United States